CLINICAL TRIAL: NCT02541123
Title: A Prospective Evaluation of Uch-l1 and Gfap Biomarker Kinetics After Mild Brain Injury Trauma
Brief Title: Evaluation of Biomarker Kinetics After Mild Brain Injury Trauma
Acronym: VIGILANT
Status: Completed | Type: Observational
Sponsor: Banyan Biomarkers, Inc (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: ATO-12
Record Dates: First submitted 2015-08-31; First posted 2015-09-04 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Head Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Craniocerebral Trauma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Cohort A: CT negative for acute intracranial lesion with initial blood draw within 4 hours of head injury
  Interventions: Other: Blood draw
- Cohort B: CT negative for acute intracranial lesion with initial blood draw within 4-6 hours of head injury
  Interventions: Other: Blood draw
- Cohort C: CT positive for acute intracranial lesion with initial blood draw within 4 hours of head injury
  Interventions: Other: Blood draw
- Cohort D: CT positive for acute intracranial lesion with initial blood draw within 4-6 hours of head injury
  Interventions: Other: Blood draw
- Cohort E: Uninjured control group
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — Initial draw followed by additional blood draws every 4 hours thereafter, up to 24 hours from the initial blood draw (not to exceed 7 blood draws). Follow up blood draw at Day 7. Control group only undergoes 2 blood draws 4 hours apart on Day 1.

SUMMARY:
The primary objective of the clinical trial is to evaluate the effect of time on levels of Ubiquitin C-terminal Hydrolase-L1 (UCH-L1) and Glial Fibrillary Acidic Protein (GFAP) biomarker levels in a population of head injured subjects over the age of 18 presenting acutely with a Glasgow Coma Scale score 13-15 as well as in a group of uninjured control subjects.

ELIGIBILITY:
Head Injured Cohorts Inclusion Criteria:

* At least 18 years of age at screening.
* Presented with a suspected traumatically induced head injury, as a result of insult to the head from an external force.
* Workup includes head CT scan, as part of clinical emergency care and CT result (CT-positive or CT-negative for acute intracranial lesions) based on the local neuroradiologist's review is available to study staff.
* CT scan and CT report used to determine eligibility must be available.
* Glasgow Coma Scale score of 13-15 at the time of Informed Consent.
* Weighs at least 110lbs (50kg), has not donated blood within the last 8 weeks, and is not anemic or has any other blood disorder which requires routine transfusions.
* First study blood sample is able to be collected into a cohort that has not been closed to enrollment
* Able to participate for up to 11 days following head injury.
* Subject or legal representative is willing to undergo the Informed Consent process prior to enrollment into this study.
* FOR CT NEGATIVE COHORTS ONLY: Subject must have experienced a Loss of Consciousness (LOC) < 30 minutes, any Alteration of Consciousness (AOC), or any Post-traumatic amnesia (PTA) following the suspected head injury AND be expected to be admitted to the hospital, or remain in hospital for at least 24 hours in order to complete Visit 1 blood draws

Head Injured Cohorts Exclusion Criteria:

* Participating in an interventional, therapeutic clinical study that may affect the results of this study (an observational study would be acceptable).
* Time of injury cannot be determined.
* Primary diagnosis of ischemic or hemorrhagic stroke.
* Venipuncture not feasible
* Neurodegenerative disease or other neurological disorder including dementia, Parkinson's disease, multiple sclerosis, seizure disorder, or brain tumors.
* History of neurosurgery within the last 30 days.
* Administration of blood transfusion after head injury and prior to the study blood draw.
* Female who is pregnant or lactating.
* Subject is otherwise determined by the Investigator to be an unsuitable candidate for participation.

Control Cohort Inclusion Criteria

* At least 18 years of age at screening
* Weighs at least 110lbs (50kg), has not donated blood within the last 8 weeks, and is not anemic or has any other blood disorder which requires routine transfusions.
* Healthy with no chronic or acute medical, neurologic, or psychiatric conditions (to the best of their knowledge).
* Able to participate for up to 5 hours following the first study blood draw.
* Willing to undergo the Informed Consent process prior to enrollment into this study.
* Subject is able to be enrolled into a control cohort that has not yet been closed to enrollment

Control Cohort Exclusion Criteria

* Participating in an interventional, therapeutic clinical study that may affect results of this study (an observational study would be acceptable).
* Subject has sustained any significant bodily injury within the past week.
* Venipuncture not feasible (i.e., skin integrity compromised at the venipuncture sites, blood vessel calcification (i.e., IV drug users, advanced atherosclerosis) both upper limbs missing (congenital or amputee)).
* Neurodegenerative disease or other neurological disorder including dementia, Parkinson's disease, multiple sclerosis, seizure disorder, or brain tumors.
* Female who is pregnant or lactating
* History of neurosurgery within the last 30 days.
* Subject is otherwise determined by the Investigator to be an unsuitable candidate for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects eligible for study participation will be over the age of 18 with a standard of care head CT result from the local neuroradiologist and be able to undergo an initial blood draw within 6 hours of head injury. Subjects who will be permitted into the study include those who will meet all the inclusion criteria and will have none of the exclusion criteria. Subjects enrolled into the control cohort will be recruited from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2016-01; Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Change in correlation of Banyan UCH-L1/GFAP Detection Assay result with acute intracranial lesions on head CT scan | initial, 4hr, 8hr,12hr,16hr, 20hr, 24hr, Day 7

CONTACTS AND LOCATIONS:
Locations (10):
- United States (7):
  - University of Florida, Gainesville, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Wayne State University, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Allegheny Singer Research Institute, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
- Klinikum rechts der Isar of the Technical University of Munich, Munich, Germany
- Hungary (2):
  - University of Pecs, Pécs
  - University of Szeged, Szeged

REFERENCES:
- [Background] Lewis LM, Papa L, Bazarian JJ, Weber A, Howard R, Welch RD. Biomarkers May Predict Unfavorable Neurological Outcome after Mild Traumatic Brain Injury. J Neurotrauma. 2020 Dec 15;37(24):2624-2631. doi: 10.1089/neu.2020.7071. Epub 2020 Sep 14. PMID 32821007